CLINICAL TRIAL: NCT06010355
Title: Breathe Easier, Philadelphia! Engaging Vulnerable Communities for Innovative Lung Cancer Care
Brief Title: Culturally Tailored Educational Video to Promote Lung Cancer Screening in Vulnerable Communities
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Study on hold pending submission of overdue annual scientific review
Sponsor: Thomas Jefferson University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Screening
Other Study IDs: iRISID-2022-1320; JT 25584 (Other: JeffTrial Number)
Record Dates: First submitted 2023-08-18; First posted 2023-08-24 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Cigarette Smoking-Related Carcinoma; Lung Carcinoma
MeSH Terms: conditions — Lung Neoplasms | interventions — Interviews as Topic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm I (Aim 1) (focus group) (Experimental): Participants participate in a focus group over 1 hour in support of the development of a culturally tailored educational video on study.
  Interventions: Procedure: Discussion
- Arm II (Aim 2) (video, interview) (Experimental): Participants watch a culturally tailored educational video over 3-5 minutes and then immediately undergo an interview in support of the refinement of a culturally tailored educational video on study.
  Interventions: Other: Media Intervention; Other: Interview
- Arm III (Aim 3) (video, test) (Experimental): Participants watch a culturally tailored educational video over 3-5 minutes and complete a brief test pre- and post-video over 30 minutes on study.
  Interventions: Other: Media Intervention; Other: Test

INTERVENTIONS:
Procedure: Discussion — Participate in focus groups
  Other Names: Discuss
  Arms: Arm I (Aim 1) (focus group)
Other: Media Intervention — Watch culturally appropriate video
  Arms: Arm II (Aim 2) (video, interview)
Other: Interview — Undergo interview
  Arms: Arm II (Aim 2) (video, interview)
Other: Media Intervention — Watch culturally appropriate video
  Arms: Arm III (Aim 3) (video, test)
Other: Test — Complete test
  Arms: Arm III (Aim 3) (video, test)

SUMMARY:
This clinical trial evaluates the impact of a culturally tailored educational video on the perceptions of lung cancer and lung cancer screening in vulnerable communities. Lung cancer is the most common cancer type. African-American communities have a higher rate than any other racial or ethnic group in the United States and accounts for the highest number of deaths among African-Americans. Lung cancer is in the top three causes of cancer death among Asian men and women. Research has shown that low-income, minority and immigrant individuals may be under resourced to make decisions about prevention programs and early detection measures for lung cancer. A culturally tailored educational video may be an effective method to help people learn about lung cancer, susceptibility toward lung cancer and lung cancer screening. This may increase lung cancer screening in vulnerable communities.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To understand barriers and opportunities for engaging three culturally distinct populations in lung cancer screening.

II. To develop three culturally tailored educational videos about lung cancer and the benefits of lung cancer screening.

III. To test the impact of the videos on susceptibility to lung cancer, knowledge of lung cancer screening, and intentions to undergo lung cancer screening in a diverse sample of at-risk individuals.

OUTLINE: Participants are assigned to 1 of 3 arms.

ARM I (AIM 1): Participants participate in a focus group over 1 hour in support of the development of a culturally tailored educational video on study.

ARM II (AIM 2): Participants watch a culturally tailored educational video over 3-5 minutes and then immediately undergo an interview in support of the refinement of a culturally tailored educational video on study.

ARM III (AIM 3): Participants watch a culturally tailored educational video over 3-5 minutes and complete a brief test pre- and post-video over 30 minutes on study.

ELIGIBILITY:
Inclusion Criteria:

* AIM 1: Participants must be African American, Korean, or Chinese adults who have either: a history of smoking, a history of lung cancer, or who have undergone lung cancer screening
* AIM 2: Participants must be African American, Korean, or Chinese adults who have either: a history of smoking, a history of lung cancer, or who have undergone lung cancer screening
* AIM 3: Those who are African American, Korean or Chinese, and are eligible for lung cancer screening, based on current screening guidelines: Current or former smokers who are between 50 and 80 years of age and who have smoked at least one pack a day for 20 years or two packs a day for 10 years

Exclusion Criteria:

* AIM 1: Those excluded from participating include children; those who are not members of the African American, Chinese, or Korean community; those who do not have one of the following: a history of smoking, a history of lung cancer, or have undergone lung cancer screening
* AIM 2: Those excluded from participating include children; those who are not members of the African American, Chinese, or Korean community; those who do not have one of the following: a history of smoking, a history of lung cancer, or have undergone lung cancer screening
* AIM 3: Those excluded from participating include children; those who are not members of the African American, Chinese, or Korean community; those who do not have a history of smoking; those who have been diagnosed with lung cancer; those who have undergone lung cancer screening in the past

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
To understand barriers and opportunities for engaging three culturally distinct populations in lung cancer screening. | From baseline to endpoint, up to 1 year
  Participants will be asked about their awareness of lung cancer screening, known or perceived barriers to screening, and potential opportunities or initiatives that could increase lung cancer screening rates in their community. Discussions will be audio recorded, transcribed by a professional transcription company, and analyzed by the study team using qualitative research methods.

SECONDARY OUTCOMES:
To develop three culturally tailored educational videos about lung cancer and the benefits of lung cancer screening | From baseline to endpoint, up to 1 year
  Ethnic cultural or other differences will be assessed and highlighted within each group, based on results from the focus groups. The beta versions of each video will be pre-tested among a small sample of individuals in each target population to refine and confirm the approach.
To test the impact of the videos on susceptibility to lung cancer, knowledge of lung cancer screening, and intentions to undergo lung cancer screening in a diverse sample of at-risk individuals. | From baseline to endpoint, up to 1 year
  First, participants will complete a brief pre-test measuring their susceptibility to lung cancer, their knowledge about lung cancer screening, their intentions to undergo lung cancer screening, and sociodemographic characteristics. Next, they will watch the video that was designed for their culture. Lastly, they will complete a post-test that includes the same measures as the pre-test, plus some additional metrics on the quality and satisfaction with the video.
  The statistical analyses will focus on describing the sociodemographic characteristics, health behaviors, and health history of participants and testing their pre-post responses for the effects of the video intervention to address Aim 3. Descriptive statistics for continuous or ordinal (e.g., Likert) scaled study variables will include means with standard deviations (or medians with first and third quartiles for skewed data) and for discrete study variables will include frequency counts with percentages.

CONTACTS AND LOCATIONS:
Overall Officials: Amy R Leader, DrPH, MPH, Principal Investigator — Thomas Jefferson University
Locations (1):
- Thomas Jefferson University Hospital, Philadelphia, Pennsylvania, United States